CLINICAL TRIAL: NCT05891717
Title: Comparative Effect of Flexibility and Resistance Training on Self-efficacy, Symptoms and Maternal Quality of Life in Postpartum Depression
Brief Title: Comparative Effect of Training on Postpartum Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0509
Record Dates: First submitted 2023-04-18; First posted 2023-06-07 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Postnatal Depression; Self Efficacy
Keywords: Strength training; Functional status; Self efficacy
MeSH Terms: conditions — Depression, Postpartum | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance training (Experimental): Group A will receive resistance training. Twice per week for 8 weeks. Total 16 sessions will given.
  Interventions: Other: Resistance training
- Flexibility training (Active Comparator): Group B will receive flexibility training. Twice per week for 8 weeks. Total 16 sessions will given.
  Interventions: Other: Flexibility training

INTERVENTIONS:
Other: Resistance training — Twice per week for 8 weeks. Total 16 sessions will given.
  Arms: Resistance training
Other: Flexibility training — Twice per week for 8 weeks. Total 16 sessions will given.
  Arms: Flexibility training

SUMMARY:
New mothers experience postpartum depression after childbirth, which commonly include mood swings, crying spells, anxiety and difficulty sleeping. Resistance training (RT) is one of the most popular methods of exercise for improving physical fitness.

This study will be a randomized clinical trial. It divide into two groups. Data will be collected from Jinnah Hospital Lahore, Family Health hospital, Johar town. Data will be taken from 36 postpartum females. Participants will be divided into 2 groups 18 women in each group: 1st group will be treated with resistance training group and 2nd group will be active comparison flexibility training group. In this study Exercises self-efficacy scale, Epidemiological studies Depression scale and MAPP-QOL (Maternal Postpartum Quality Life Questionnaire) will be used as subjective measurements.

DETAILED DESCRIPTION:
New mothers experience postpartum depression after childbirth, which commonly include mood swings, crying spells, anxiety and difficulty sleeping. Postpartum depression typically begins within the first two to three days after delivery and may last for up to several weeks or months. Activity and mobility are an integral part of human life that is manifested in a special way in each period. Postpartum life has caused lack of movement, the risk factor of depression and difficulty in maternal life. Resistance training (RT) is one of the most popular methods of exercise for improving physical fitness. A logical approach to treatment, therefore, would be to improve postpartum life. Flexibility exercises are not just for gymnasts, but rather for everyone. Along with the better range of motion, it decreases risks of injuries, increases blood supply and nutrients to joints, reduces muscular tension and help to improve quality of life.

This study will be a randomized clinical trial. Subjects meeting the predetermined inclusion and exclusion criteria will divide into two groups. Data will be collected from Jinnah Hospital Lahore, Family Health hospital, Johar town. After informed consents were obtained, data will collect. After taking written consent from participants who meet the inclusion criteria, data will be taken from 36 postpartum females. Participants will be divided into 2 groups 18 women in each group: 1st group will be treated with resistance training group and 2nd group will be active comparison flexibility training group. Pre-treatment assessment and Post treatment reading will be done using Exercises self-efficacy scale, Epidemiological studies Depression scale and MAPP-QOL (Maternal Postpartum Quality Life Questionnaire) as subjective measurements. Recorded values will be analyzed for any change using SPSs version 25.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 40
* 6 weeks to 8 months postpartum females
* primiparous or multiparous postnatal wome

Exclusion Criteria:

* Family history of depression
* Hospitalization for a psychiatric disorder in the past 6 months; and currently receiving antidepressant medication or psychotherapy for depression.
* Pregnant women
* Women with psychiatric diagnoses other than depression

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum Female
Enrollment: 36 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Exercise self efficacy | 8 weeks
  A 9-item questionnaire that focuses on the self-efficacy expectations for exercise for older adults; specifically the ability to continue to exercise despite barriers. The participant is asked about their confidence level, on a scale from 0 (not confident) to 10 (very confident)
Epidemiological studies Depression scale | 8 weeks
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a brief self-report questionnaire developed in 1977 by Laurie Radloff to measure depressive symptoms severity in the general population
MAPP-QOL ( Maternal Postpartum Quality Life Questionnaire) | 8 weeks
  Maternal Postpartum Quality of Life (MAPP-QOL) questionnaire, which is a self-administered instrument that measures quality of life during the early postnatal period. 12 The MAPP-QOL is composed of five domains and demonstrates convergent validity with measures of life satisfaction and mood states.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phill, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posmontier B. Functional status outcomes in mothers with and without postpartum depression. J Midwifery Womens Health. 2008 Jul-Aug;53(4):310-8. doi: 10.1016/j.jmwh.2008.02.016. PMID 18586183
- [Background] Papamarkou M, Sarafis P, Kaite CP, Malliarou M, Tsounis A, Niakas D. Investigation of the association between quality of life and depressive symptoms during postpartum period: a correlational study. BMC Womens Health. 2017 Nov 21;17(1):115. doi: 10.1186/s12905-017-0473-0. PMID 29162087
- [Background] Fragala MS, Cadore EL, Dorgo S, Izquierdo M, Kraemer WJ, Peterson MD, Ryan ED. Resistance Training for Older Adults: Position Statement From the National Strength and Conditioning Association. J Strength Cond Res. 2019 Aug;33(8):2019-2052. doi: 10.1519/JSC.0000000000003230. PMID 31343601
- [Background] Hooker QL, Lanier VM, Roles K, van Dillen LR. Motor skill training versus strength and flexibility exercise in people with chronic low back pain: Preplanned analysis of effects on kinematics during a functional activity. Clin Biomech (Bristol). 2022 Feb;92:105570. doi: 10.1016/j.clinbiomech.2021.105570. Epub 2022 Jan 3. PMID 35045374
- [Background] Mirghafourvand M, Bagherinia M. Relationship between maternal self-efficacy and functional status four months after delivery in Iranian primiparous women. J Psychosom Obstet Gynaecol. 2018 Dec;39(4):321-328. doi: 10.1080/0167482X.2017.1394290. Epub 2017 Nov 2. PMID 29094655